CLINICAL TRIAL: NCT02292043
Title: Effects of HTEA ON Heart Failure Secondary to Idiopathic Dilated Cardiomyopathy or Post-myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Wei Liu, Prof. Liu, Harbin Medical University
Other Study IDs: wei liu
Record Dates: First submitted 2014-10-31; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- idiopathic dilated cardiomyopathy group: idiopathic dilated cardiomyopathy group treated with HTEA
  Interventions: Drug: HTEA
- post-myocardial infarction group: post-myocardial infarction group treated with TEA
  Interventions: Drug: HTEA

INTERVENTIONS:
Drug: HTEA — HTEA

SUMMARY:
The investigators would evaluate the effects of the novel method, HTEA on cardiac function in the heart failure patients secondary to idiopathic dilated cardiomyopathy and post-myocardial infarction.

DETAILED DESCRIPTION:
The investigators would evaluate the effects of the novel method, HTEA on cardiac function in the heart failure patients secondary to idiopathic dilated cardiomyopathy and post-myocardial infarction. The specific index is 6 miniutes walk distance, echocardiography, NYHA, NTproBNP level, peripherial WBC, RBC, PLT, Cre, UA, K+, Na+ upon entrance to hospital and 4 weeks after HTEA treatment, and 3 months after discharge. The morbidity and re-hospitalization would also calculated 3 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* 90 chronic cardiac failure patients in our hospital were selected and divided into two groups.

Exclusion Criteria:

* Vavular diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heart failure.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Morbidity | 1 months to 3 months after discharge

SECONDARY OUTCOMES:
The decreased degree of NT-proBNP higher than 30% | 3 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: wei liu, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (2):
- China (2):
  - Ren Xiaohui, Harbin, Heilongjiang
  - the first affiliated hospital of Harbin Medical University, Harbin, Heilongjiang